CLINICAL TRIAL: NCT01648803
Title: Wearable Movement Sensors for Assessing Motor Impairments and Dyskinesias in Parkinson Disease
Acronym: APDMclinic
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: RSRB39530
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to measure motor fluctuations and dyskinesias in patients with Parkinson's disease using movement sensors (accelerometers and gyroscopes) to determine if this is a feasible measure to use in addition to self report, and eventually the goal will be to replace self report with a more reliable measure such as movement sensors.

DETAILED DESCRIPTION:
Patients with Parkinson disease and motor fluctuations will wear movement sensors during their regular clinic visit with the principal investigator. The visit will be videotaped and medication status (ON without dyskinesia, ON with dyskinesia, or OFF) will be independently rated from review of the video.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will be included in the study have probable or definite idiopathic PD (CAPSIT criteria (23)), Hoehn & Yahr stage 2-4;
* One or more of the following PD-associated motor impairments experienced in the week prior to enrollment (based on history and/or examination): motor fluctuations (end of dose wearing off with hypokinesia and/or levodopa-induced choreiform dyskinesias), tremor, freezing of gait, or frequent falls (≥ 1 per week).

Exclusion Criteria:

* Neurological disorders (other than PD) or orthopedic deficits that, in the investigator's judgement, contribute substantially to impaired movement (e.g. stroke with motor sequelae;
* Essential tremor;
* Severe osteoarthritis);
* Cognitive impairment sufficiently severe to interfere with informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial study population for this pilot study will consist of approximately 20 people. The study will be comprised of approximately equal numbers of men and women. The gender and ethnic origins of the patients seen in the University of Rochester Movement Disorders Center (from which subjects will be recruited) are approximately 60% male and 40% female; 91% Caucasian, 1% African American, 1% Hispanic, and 0.5% Asian (6% Unknown). There are no restrictions on gender or race, however non-english speaking patients will be excluded as the consent form will initially only be available in English. Parkinson disease is exceedingly rare in children and only adults will be enrolled for this study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
1-3Hz gyroscope signal power | 30 second windows spanning the observation period

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Burack, MD PhD, Principal Investigator — University of Rochester Medical Center Dept. of Neurology
Locations (1):
- University of Rochester, Rochester, New York, United States